CLINICAL TRIAL: NCT00311896
Title: Multicentric, Randomized, Placebo Controlled and Double-blind Study to Evaluate the Efficacy and Safety of Antithrombotic Prophylaxis With Bemiparin (3,500 UI/Day) in Cancer Patients With a Central Venous Catheter (CVC)(BECAT)
Brief Title: Efficacy & Safety of Prophylaxis With Bemiparin in Cancer Patients With a Central Venous Catheter (BECAT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor stopped due to difficulties to recruit 402 patients required by protocol
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Laboratorio farmacéutico ROVI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ICT-BEM-2004-02; BECAT
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Cancer; Thrombosis
Keywords: Cancer; Thrombosis; Catheter; Bemiparin; Prophylaxis
MeSH Terms: conditions — Neoplasms; Thrombosis | interventions — bemiparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bemiparin (Experimental)
  Interventions: Drug: Bemiparin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bemiparin
  Arms: Bemiparin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the subcutaneous administration for 45 days of Bemiparin (3,500 UI/day) in cancer patients with a CVC, to prevent CVC-related deep venous thrombosis (CVC-DVT)

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a common complication in patients with cancer principally in association with central vein catheters (CVC). The clinical benefit of antithrombotic prophylaxis for CVC-related VTE in cancer patients remains unclear.The aim of this study is to evaluate the efficacy and safety of the administration of Bemiparin in cancer patients with a central venous catheter (CVC). This study is designed as a multicenter, randomized, double-blind, placebo-controlled study. On the day of CVC insertion, eligible patients are randomly assigned to receive subcutaneously either bemiparin (3,500 UI/day) or placebo by using preloaded syringes for 45 days.

The primary efficacy endpoint will be the combined incidence during the double blind treatment period of Clinical or symptomatic CVC-DVT verified objectively (Doppler ultrasonography or phlebography)and subclinical or asymptomatic CVC-DVT confirmed by elective bilateral Doppler ultrasonography performed 45±5 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old of either sex who have given their informed consent to participate in the study.
* Patients with a neoplastic process, with a CVC for the administration of anti-tumoral treatment or any other treatment related to the neoplastic process.
* Patients with a platelet count above 30,000/mm3.
* Patients with no hemorrhagic symptomatology at the time of their inclusion

Exclusion Criteria:

* Patients with a history of clinically evident hemorrhagic episodes and/or with increased bleeding due to any other homeostatic alteration that contraindicates anticoagulant treatment and/or in the past two months have presented at least one of the following: active hemorrhaging or organic lesions susceptible to bleeding (e.g. active peptic ulcer, hemorrhagic cerebrovascular accident, aneurysms).
* Major surgery in the past two months.
* Known hypersensitivity to LMWH, heparin or substances of porcine origin.
* Patients with congenital or acquired bleeding diathesis.
* Damage to or surgical interventions of the central nervous system, eyes and ears within the past 6 months.
* Acute bacterial endocarditis or slow endocarditis.
* Patients with a history of heparin-associated thrombocytopenia.
* Patients with severe renal failure (serum creatinine over 2 mg/dl) or hepatic insufficiency (with values of AST and/or ALT > 5 times the normal value established by the reference range of the local hospital laboratory).
* Severe arterial hypertension (systolic blood pressure over 200 mmHg and/or diastolic blood pressure over 120 mmHg).
* Patients with suspected inability/or inability to comply with treatment and/or complete the study.
* Patients who are participating in another clinical trial or have done so in the past 30 days.
* Patients with a life expectancy less than 3 months.
* Women who are pregnant or breast-feeding, or with the possibility of becoming pregnant during the study.
* Patients on treatment with anticoagulants or who have been on treatment during the week previous to insert the CVC (including prophylaxis with heparin for hepatic veno-occlusive disease).
* Patients diagnosed with acute leukemia or awaiting a transplant from hematopoietic progenitors during the 90 days of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2005-07; Primary Completion 2009-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical or symptomatic CVC-DVT verified objectively (Doppler ultrasonography or phlebography).
Subclinical or asymptomatic CVC-DVT confirmed by elective bilateral Doppler ultrasonography performed 45±5 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Rocha, MD, Study Chair — Clinica Universitaria de Navarra; Ramon Lecumberri, MD, Principal Investigator — Clinica Universitaria de Navarra; Vicente Vicente, MD, Principal Investigator — Hospital Morales Meseguer; Pascual Marco, MD, Principal Investigator — Hospital General Universitario de Alicante; José Mateo, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Albert Font, MD, Principal Investigator — Germans Trias i Pujol Hospital; Carmen Arratibel, MD, Principal Investigator — Complejo Hospitalario de Donostia; Francisco J. Capote, MD, Principal Investigator — Hospital Universitario Puerta del Mar; Miguel Angel De gregorio Ariza, MD, Principal Investigator — Hospital Clinico Universitario Lozano Blesa-Zaragoza; Isabel Picón Roig, MD, Principal Investigator — Instituto Valenciano de Oncología; Ricardo González Del Val Subirats, MD, Principal Investigator — Hospital General Universitario Gregorio Marañón; Carlos Bosh Roig, MD, Principal Investigator — Hospital Universitario Doctor Peset; Pedro Pérez-Segura, MD, Principal Investigator — Hospital Clínico San Carlos-Madrid.; Vicente Alberola, MD, Principal Investigator — Hospital Arnau de Vilanova de Valencia; César Rodríguez Sánchez, MD, Principal Investigator — Hospital Clínico de Salamanca; Ignacio Alberca Silva, MD, Principal Investigator — Hospital Clínico de Salamanca; Javier García Frade, MD, Principal Investigator — Hospital del Rio Hortega; Carmen Sedano, MD, Principal Investigator — Hospital Marqués de Valdecilla; Natividad Gómez, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Amalia Velasco, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Carmen Rodríguez Pinto, MD, Principal Investigator — Hospital Universitario Central de Asturias; Mihai Ciochinaru, MD, Principal Investigator — Cenral Emergency Clinical Military H.; Cornelia Toganel, MD, Principal Investigator — District Emergency Clinical Hospital; Csaba Bela Szekely, MD, Principal Investigator — Arad District Hospital; Mihaela Danciulescu, MD, Principal Investigator — Filantropia District Hospital; Constantin Volovat, MD, Principal Investigator — Oncology Medical Center Iasi; Mircea Cazacu, Prof., Principal Investigator — University "CF" Clinical Hospital; Eliade Ciuleanu, MD, Principal Investigator — Oncology Institute Cuj-Napoca; Florin Bacanu, md, Principal Investigator — Sf Maria Clinical Hospital
Locations (19):
- Romania (8):
  - Arad County Hospital, Arad
  - Cenral Emergency Clinical Military H., Bucharest
  - Sf Maria Clinical Hospital, Bucharest
  - Oncology Institute Cuj-Napoca, Cluj-Napoca
  - University "CF" Clinical Hospital, Cluj-Napoca
  - Filantropia District Hospital, Craiova
  - Oncology Medical Center, Iasi, Iași
  - District Emergency Clinical Hospital, Târgu Mureş
- Spain (11):
  - Hospital General de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Complejo Hospitalario de Donostia, Donostia / San Sebastian
  - Hospital Clínico San Carlos-Madrid., Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Morales Meseguer, Murcia
  - Clínica Universitaria de Navarra, Pamplona
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza